CLINICAL TRIAL: NCT00707915
Title: Effects of Discontinuation of Benzodiazepine-derivative Hypnotics on Cognitive and Motor Functions in Elderly Persons: a Pilot Study
Brief Title: Effects of Discontinuation of Benzodiazepine-derivative Hypnotics on Cognitive and Motor Functions in Elderly Persons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minamihanno Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH0001
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Adverse Effects
Keywords: aged; benzodiazepines; hypnotics; cognition; posture
MeSH Terms: interventions — Benzodiazepines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose reduction (Experimental): The benzodiazepine dose will be discontinued in 4 weeks by a weekly 25% reduction. Participants will be observed for 8 weeks.
  Interventions: Drug: Drug: Benzodiazepine (listed out below)

INTERVENTIONS:
Drug: Drug: Benzodiazepine (listed out below) — The benzodiazepine (BZD) dose will be discontinued in 4 weeks by a weekly 25% reduction. BZD-derivative hypnotics will include brotizolam, flunitrazepam, etizolam, quazepam, estazolam, nitrazepam, flurazepam, and diazepam.
  All psychotropic agents other than the BZD-derivative hypnotics will be kept constant throughout the study. In addition, the use of trazodone (25-100 mg/day) will be allowed anytime throughout the study period. Subjects will be observed for 8 weeks.

SUMMARY:
Benzodiazepines (BZDs) have been reported to cause negative impacts on motor as well as cognitive functions, which in turn could result in lethal incidents including falls especially in the elderly. This notwithstanding, few trials have evaluated a feasibility and benefits of discontinuing BZD-derivative hypnotics in a systematic manner in this frail population. In this 8-week open-label study, we examined changes in motor and cognitive functions following the discontinuation of BZD hypnotics in older persons.

OBJECTIVES & HYPOTHESES

1. Primary Objective The primary objective is to examine the feasibility of discontinuing BZD-derivative hypnotics in older people.
2. Secondary Objectives

   1. One of the secondary objectives is to examine the magnitude of discontinuing BZD-derivative hypnotics in the stability of body.
   2. Another secondary objective is to examine the magnitude of discontinuing BZD-derivative hypnotics in cognitive function.

Hypotheses

1. More than 80% of the participants will complete and tolerate all the study procedures.

2a. Participants will show an improvement in the stability of body. 2b. Participants will show an improvement in the cognitive function globally as well as specifically in attention.

DETAILED DESCRIPTION:
Benzodiazepines (BZDs) have been reported to cause negative impacts on motor as well as cognitive functions, which in turn could result in lethal incidents including falls especially in the elderly. This notwithstanding, few trials have evaluated a feasibility and benefits of discontinuing BZD-derivative hypnotics in a systematic manner in this frail population. In this study, we examined changes in motor and cognitive functions following the discontinuation of BZD hypnotics in older persons.

In this 8-week open-label study, subjects aged 50 or older who receive BZD as a hypnotic and do not have any unstable physical illness, or neurological disorder will be recruited. The BZD dose will be discontinued in 4 weeks by a weekly 25% reduction.

Following assessments will be performed at baseline 12 hours postdose and at endpoint: the Clinical Stabilometric Platform (CSP), the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and the Critical Flicker Fusion Test (CFF), the Leeds Sleep Evaluation Questionnaire (LSEQ). The CSP measures the stability of body, with the eyes opened or closed.

All psychotropic agents other than the BZD-derivative hypnotics will be kept constant throughout the study.

The dose reduction will be terminated if any of the following conditions are fulfilled:

1. Clinical worsening in sleep defined as a CGI-Global Improvement score of 7
2. Participant's request
3. Clinical decision on the part of the physician of record or independent consulting physician In the event that a participant needs a dose increment for anxiety and insomnia, the dose will be increased back to the previous dose, and they will be followed for the rest of the study period. In addition, the use of trazodone (25-100 mg/day) will be allowed anytime throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of any race or ethnicity with any psychiatric diagnosis
* Age of 50 and older
* Having been treated with an BZD-derivative hypnotic drug at a steady dose for at least 4 weeks

Exclusion Criteria:

* Incapacity to follow the instructions.
* Unstable physical illness or significant neurological disorder
* Psychiatric concerns raised by the physician of record regarding participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Tsunoda, MD, Principal Investigator — Minamihanno Hospital
Locations (1):
- Minamihanno Hospital, Hannou, Saitama, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: psychiatric hospital & nursing home
Groups:
- Dose-reduction: The benzodiazepine dose will be discontinued in 4 weeks by a weekly 25% reduction. Participants will be observed for 8 weeks.
Period: Overall Study
Arm/Group | Dose-reduction
Started | 30
Effects of Discontinuing Benzodiazepine | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose-reduction
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 79.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  Japan | 30

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate
Description: The number of subjects who have successfully completed dose-reduction and all the assessments scheduled until week 8 divided by the total number of enrolled subjects
Time Frame: 8 weeks
Measure: Number; unit: percentage of successful completers
Arm/Group | Dose-reduction
Number analyzed (Participants) | 30
percentage of successful completers | 26

2. Secondary Outcome: A Change in a Total Scale Score in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Japanese Version, From Baseline to Week 8.
Description: This brief test is to assess areas of cognitive functioning and profile impairment across domains with 12 subtests, including: List Learning, Story Memory, Figure Copy, Line Orientation, Digit Span, Coding, Picture Naming, Semantic Fluency, List Recall, List Recognition, Story Recall, and Figure Recall. This assessment is repeatable and not subject to practice effects. A total scale score ranges between 40 and 160; a higher score indicates better cognitive function. A change in the score between the baseline and week 8 is defined as a secondary outcome measure.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose-reduction
Number analyzed (Participants) | 26
units on a scale | 8.8 (3.2)

3. Secondary Outcome: Clinical Stabilometric Platform (CSP)
Description: CSP (ANIMA® GS-7, Tokyo) measures a total length of the trunk motion by varying the resistance applied to the platform for 30 seconds with eyes closed with feet together. Change in the total length of the trunk motion from baseline to week 8 will be recorded.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dose-reduction
Number analyzed (Participants) | 26
cm | -1.5 (0.8)

4. Secondary Outcome: Critical Flicker Fusion Test (CFF)
Description: The CFF threshold has been regarded as a functional measure of psychomotor function. Sub-threshold intermittent light is perceived as a flicker. If the frequency is gradually increased, the flicker becomes gradually less distinct until it is finally perceived as a continuous light (fusion threshold). The device (T.K.K.501c) provides luminance with a mean intensity of 500Lux±10% and a range of frequency of 20-60Hz. A change in the critical fusion frequency from baseline to week 8 will be recorded.
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Dose-reduction
Number analyzed (Participants) | 26
Hz | 2.1 (1.5)

5. Secondary Outcome: Leeds Sleep Evaluation Questionnaire (LSEQ)
Description: The LSEQ comprises 10 self-rating 100-mm-line analogue questions regarding changes in the quality of sleep and early morning behavior, following any given intervention. Scores range between 0 and 100. Scores beneath 50 indicate better sleep. This will be performed at week 8.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose-reduction
Number analyzed (Participants) | 26
units on a scale | 46.4 (32.9)

6. Secondary Outcome: Clinical Global Impression (CGI)
Description: The CGI rating scales are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders (Guy, W., 1976). The CGI - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. This will be performed at week 8.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose-reduction
Number analyzed (Participants) | 30
units on a scale | 4.2 (1.8)

ADVERSE EVENTS:
Arm/Group | Dose-reduction
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No